CLINICAL TRIAL: NCT03021837
Title: The Effect of Steroids for Fetal Lung Maturity on Maternal Glucose Levels
Brief Title: The Effect of Steroids on Maternal Glucose Levels
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Dorothea Mostello, MD, Principal Investigator, St. Louis University
Other Study IDs: 21014a; NCT02912091 (obsolete NCT alias)
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all patients: Patient receiving antenatal corticosteroid course for fetal lung maturity consisting of betamethasone or dexamethasone Women without known gestational diabetes and women with non-insulin requiring gestational diabetes (A1GDM)
  Interventions: Other: antenatal corticosteroid

INTERVENTIONS:
Other: antenatal corticosteroid — Will look at maternal glucose level after corticosteroids

SUMMARY:
This study will look at blood sugar levels in pregnant women who have been given a glucocorticoid (steroid) medication to enhance fetal lung maturity. The findings will help determine the likelihood, predictive value, adverse effects, response of patients diagnosed with gestational diabetes and time course of blood sugar elevation following steroids.

DETAILED DESCRIPTION:
Few studies have examined the effects on maternal glucose levels from corticosteroids, which are given during some complicated pregnancies to enhance fetal lung maturity when early delivery is expected. The applicability of these studies is limited by the presence of confounding factors and low numbers of participants (ranging between 7 and 50). Two relevant studies are by Mastrobiattista at al and Gurbuz et al. These studies had 7 and 40 subjects respectively, and studied the change in maternal 1-hour glucose tolerance tests following administration of steroids for fetal lung maturity. The 1-hour tests involve a standard oral glucose challenge and are used to screen for gestational diabetes; thus, they may not reflect the changes in circulating glucose levels from typical sources of glucose (such as meals) anticipated with steroid administration. Both studies showed a change in the results of glucose tolerance testing and concluded that screening for gestational diabetes should be delayed at least 72 hours to 1 week after completion of the steroid course. Neither study looked at maternal glucose values within the first 48 hours of giving the first dose of steroids, and neither addressed whether diabetes could be diagnosed alternatively by the maternal glucose response within the first 48 hours following steroid administration.

It has been the investigator's clinical observation that glucose values may be highest during those first 48 hours. Another study looked at the effect of various doses of insulin on the degree of hyperglycemia for the first 3 days following steroid administration and showed increases in glucose values even in the insulin-treated. Unfortunately, some subjects in that study had concurrent treatment with another agent known to cause hyperglycemia.

No standards of care exist to guide whether to monitor glucose values after steroid administration for fetal lung maturity. The time course of glucose elevations is not clear, and how often the glucose elevations reach a level that would generally warrant treatment is unknown. When glucose monitoring is performed, no standard exists to guide the duration or frequency of monitoring.

Detecting maternal hyperglycemia is important for several reasons, including:

1. High maternal glucose levels lead to high fetal levels and prompt a fetal response to the high glucose levels. Some of the pregnancies may go on to deliver while the maternal glucose levels are still high, resulting in a higher risk of neonatal hypoglycemia in the nursery and an increased risk of acidosis and injury in the brain if periods of distress occur during labor. By the nature of the clinical situations, most fetuses born in the first few days following administration of steroids will also be preterm and possibly already have additional factors which put them at risk for complications in labor and the nursery, so the hyperglycemia compounds the risk for them.
2. The maternal hyperglycemia may complicate the maternal course at a time when the pregnant woman is receiving other medications to control her premature labor or obstetric condition that prompted the use of the steroids in the first place. Fluid balance and constitutional symptoms may be affected by high glucose values. Rarely, diabetic ketoacidosis may be precipitated in someone with no history of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine pregnancy at 22 weeks to 36 weeks gestation at time of steroid administration
* Singleton
* Patient receiving antenatal corticosteroid course for fetal lung maturity consisting of betamethasone or dexamethasone
* Age range: 14yo-50yo
* Women without known gestational diabetes and women with non-insulin requiring gestational diabetes (A1GDM)

Exclusion Criteria:

* Women with known gestational diabetes (diagnosed before steroid administration) that has required insulin or other medical therapy to control
* Women with overt diabetes which predates pregnancy.
* Chronic terbutaline therapy or other concurrent chronic beta-adrenergic agonist use
* Patients on parenteral or oral corticosteroids for reasons other than to improve fetal lung maturity
* Multiple gestation

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant patients, who meet Inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-08-24 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2015-03-17 (Actual)

PRIMARY OUTCOMES:
The length of time that maternal glucose levels remain elevated after steroid administration. | 6 hours
  Time until glucose levels return to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea Mostello, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No